CLINICAL TRIAL: NCT03245372
Title: Goal Directed Therapy Versus Standard Care in Lung Resection Surgery, a Randomized, Controlled Trial (GDT-thorax Study).
Brief Title: Goal Directed Therapy Versus Standard Care in Lung Resection Surgery (GDT-thorax Study).
Acronym: GDT-thorax
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2017/118
Record Dates: First submitted 2017-07-17; First posted 2017-08-10 (Actual); Results first posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Goal Directed Therapy; Fluid Therapy
Keywords: cardiac output; perioperative care; postoperative complications
MeSH Terms: conditions — Postoperative Complications | interventions — Standard of Care; Early Goal-Directed Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard care (Active Comparator): Basic intraoperative hemodynamic objectives
  Interventions: Procedure: Standard care
- Goal directed therapy (Experimental): Target value is a cardiac index equal or superior to 2.2 l/min/m2.
  Interventions: Procedure: Goal directed therapy

INTERVENTIONS:
Procedure: Standard care — Heart rate 60-100 beats per minute, mean arterial pressure 65 mm Hg, serum lactate 2 mmol/L, oxygen saturation 95 % (90 % during one lung ventilation).
  Other Names: Conventional fluid and hemodynamic management
  Arms: Standard care
Procedure: Goal directed therapy — The hemodynamic algorithm will be based on systolic volume index and fluid challenges. FloTrac sensor (this sensor connects to any existing arterial catheter and provides advanced hemodynamic parameters through pulse contour analysis) and EV1000 clinical platform (clinical platform from Edwards Lifesciences that provides advanced hemodynamic monitoring) will be used to calculate cardiac index and systolic volume index.
  Other Names: Goal directed fluid and hemodynamic management
  Arms: Goal directed therapy

SUMMARY:
The primary aim of this study is to quantify and compare the hemodynamic control of cardiac index in patients who receive either goal-directed therapy or standard hemodynamic management in lung resection surgery

DETAILED DESCRIPTION:
The investigators hypothesize that the percentage of the intraoperative time in which the cardiac index is equal or superior to 2.2 l/min/m2 is higher in goal directed therapy

ELIGIBILITY:
Inclusion Criteria:

* Adults patients ( 18 years old)
* Written informed consent
* Elective lung resection surgery (open or thoracoscopic lung lobectomy)

Exclusion Criteria:

* Severe obesity
* Moderate to severe aortic insufficiency
* Renal failure requiring hemodialysis
* Left ventricle ejection fraction less than 35 %
* Urgent surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Bertomeu, MD-PhD, Study Chair — Andaluz Health Service
Locations (1):
- University hospital Virgen del Rocío, Seville, Spain

IPD SHARING:
Plan to Share IPD: Yes
Yes. Anonymized data for individual patient data is planned to be shared with all participants within 6 months of data completion
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 6 months after the completion of data analysis
Access Criteria: colaborators in the investigation will be open to the whole data base and analysis performed

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 31 patients signed informed consent, but there was a pre-randomization exclusion (a patient was selected and signed informed consent) because surgeons decided to carry out a less aggressive surgery from the start (atypical lung resection instead of lobectomy). That happened in only one case.
Period: Overall Study
Arm/Group | Standard Care | Goal Directed Therapy
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Goal Directed Therapy | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (9.91) | 67.33 (8.64) | 67.37 (9.137)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 11 | 13 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 15 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 15 | 15 | 30
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.96 (4.35) | 24.64 (3.39) | 25.3 (3.89)
Smoking history [Count of Participants; unit: Participants] | 12 | 13 | 25
Smoking exposure [Median (Standard Deviation); unit: pack-years] | 33.79 (31.27) | 34.07 (20.15) | 33.93 (25.85)
ASA Physical Status Classification System [Count of Participants; unit: Participants] — The ASA Physical Status Classification System has been in use for over 60 years. The purpose of the system is to assess and communicate a patient's pre-anesthesia medical co-morbidities. It can be helpful in predicting perioperative risks.
  * ASA I: A normal healthy patient
  * ASA II: A patient with mild systemic disease
  * ASA III: A patient with severe systemic disease
  * ASA IV: A patient with severe systemic disease that is a constant threat to life.
  * ASA V: A moribund patient who is not expected to survive without the operation
  ASA III-IV-V may have worse outcomes than I or II
  Participants
    ASA II | 3 | 8 | 11
    ASA III | 12 | 7 | 19
Hypertension [Count of Participants; unit: Participants] | 9 | 11 | 20
Dyslipidemia [Count of Participants; unit: Participants] | 9 | 7 | 16
Diabetes Mellitus [Count of Participants; unit: Participants] | 3 | 4 | 7
Ischemic heart disease [Count of Participants; unit: Participants] | 0 | 3 | 3
Atrial fibrillation [Count of Participants; unit: Participants] | 2 | 1 | 3
Chronic kidney disease [Count of Participants; unit: Participants] | 2 | 3 | 5
COPD grade GOLD is equal or superior to 2 [Count of Participants; unit: Participants] — COPD (chronic obstructive pulmonary disease) stages and the GOLD (Global Initiative for Obstructive Lung Disease) criteria:
  * Stage I (Early)
  * Stage II (Moderate)
  * Stage III (Severe)
  * Stage IV (Very Severe)
  COPD grade II or above II may have worse outcomes than patients grade I or without that desease
  Participants | 2 | 3 | 5
cerebrovascular disease [Count of Participants; unit: Participants] | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of the Intraoperative Time in Which the Cardiac Index is Equal or Superior to 2.2 l/Min/m2 (%)
Description: To compare the degree of hemodynamic control of cardiac index in both groups: Percentage of the intraoperative time in which the cardiac index is equal or superior to 2.2 l/min/m2.
Time Frame: During the total duration of the surgery, on average 4 hours. We include the time from the start of maintenance of general anesthesia to the moment of extubation of the patient.
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Standard Care | Goal Directed Therapy
Number analyzed (Participants) | 15 | 15
percentage of time | 97 [92 to 99] | 91 [79 to 98]
Statistical Analysis 1: Comparison: Standard Care vs Goal Directed Therapy; Test type: Superiority; p = 0.114, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Tissue Perfusion Marker: Lactate
Description: To compare lactate in the first 24 hours in both groups
Time Frame: Within 24 hours after lung surgery
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Standard Care | Goal Directed Therapy
Number analyzed (Participants) | 15 | 15
mmol/L | 0.70 [0.5 to 1.20] | 0.80 [0.6 to 1]
Statistical Analysis 1: Comparison: Standard Care vs Goal Directed Therapy; Test type: Superiority; p = 0.692, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Tissue Perfusion Marker: SvcO2
Description: To compare SvcO2 (central venous oxygen saturation) in the first 24 hours in both groups
Time Frame: Within 24 hours after lung surgery
Measure: Mean (Standard Deviation); unit: percentage of saturation
Arm/Group | Standard Care | Goal Directed Therapy
Number analyzed (Participants) | 15 | 15
percentage of saturation | 66.03 (7.16) | 70.16 (5.14)
Statistical Analysis 1: Comparison: Standard Care vs Goal Directed Therapy; Test type: Superiority; p = 0.082, t-test, 2 sided

4. Secondary Outcome: Oxygenation Marker: PaO2/FiO2 Ratio
Description: To compare PaO2/FiO2 ratio (ratio of arterial oxygen partial pressure to fractional inspired oxygen) in the first 24 hours in both groups
Time Frame: Within 24 hours after lung surgery
Measure: Median (Inter-Quartile Range); unit: mm Hg
Arm/Group | Standard Care | Goal Directed Therapy
Number analyzed (Participants) | 15 | 15
mm Hg | 331.43 [286.66 to 398.09] | 339.05 [301.43 to 390.47]
Statistical Analysis 1: Comparison: Standard Care vs Goal Directed Therapy; Test type: Superiority; p = 0.443, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Fluid Balance
Description: To compare fluid balance (differences between the amount of water taken into the body and the amount excreted or lost) in the first 24 hours in both groups
Time Frame: After 24 hours of finalization of lung surgery
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Standard Care | Goal Directed Therapy
Number analyzed (Participants) | 15 | 15
milliliters | 647.17 (700.57) | 748.83 (579.46)
Statistical Analysis 1: Comparison: Standard Care vs Goal Directed Therapy; Test type: Superiority; p = 0.668, t-test, 2 sided

6. Secondary Outcome: Observation of Acute Kidney Injury (AKI)
Description: To compare the Number of Participants with Acute Kidney Injury in both groups
Time Frame: After 72 hours of finalization of lung surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Goal Directed Therapy
Number analyzed (Participants) | 15 | 15
Participants | 3 | 5
Statistical Analysis 1: Comparison: Standard Care vs Goal Directed Therapy; Test type: Superiority; p = 0.516, Chi-squared

7. Secondary Outcome: Observation of Acute Respiratory Distress Syndrome (ARDS)
Description: To compare the he Number of Participants with Acute Respiratory Distress Syndrome in both groups
Time Frame: Within 30 days after lung surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Goal Directed Therapy
Number analyzed (Participants) | 15 | 15
Participants | 0 | 0

8. Secondary Outcome: Duration of Hospital Stay
Description: To compare hospital stay in both groups
Time Frame: Within 30 days after lung surgery
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard Care | Goal Directed Therapy
Number analyzed (Participants) | 15 | 15
days | 4 [4 to 5] | 5 [4 to 6]
Statistical Analysis 1: Comparison: Standard Care vs Goal Directed Therapy; Test type: Superiority; p = 0.229, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Mortality
Description: To compare the mortality rate in both groups
Time Frame: Within 30 days after lung surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Goal Directed Therapy
Number analyzed (Participants) | 15 | 15
Participants | 1 | 0
Statistical Analysis 1: Comparison: Standard Care vs Goal Directed Therapy; Test type: Superiority; p = 1, Fisher Exact

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Standard Care | Goal Directed Therapy
All-Cause Mortality (participants affected / at risk) | 1/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 3/15 | 4/15
Other Adverse Events (participants affected / at risk) | 12/15 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=15) | Goal Directed Therapy (N=15)
Acute Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Thoracic Pain (Cardiac disorders) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atrial Fibrillation Paroxysmal (Cardiac disorders) | 1 (1) | 1 (1)
Severe Subcutaneous Emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=15) | Goal Directed Therapy (N=15)
Acute Kidney Injury (Renal and urinary disorders) | 3 (3) | 5 (5)
Exanthema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Postoperative Nausea and Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (4)
Surgical Site Infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arterial Hypotension (Cardiac disorders) | 4 (4) | 9 (9)
Fever (General disorders) | 1 (1) | 0 (0)
Mild-Moderate Subcutaneous Emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
This is a pilot study and the clinician (anesthesiologist) who performed the anesthetic procedure had to know the assignment of the arm. The intervention was limited to the intraoperative period. Postoperative morbidity and mortality surveillance was limited to one month. The study, therefore, was not designed to have sufficient power to detect significant differences in major postoperative complications.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-29): https://cdn.clinicaltrials.gov/large-docs/72/NCT03245372/Prot_SAP_001.pdf